CLINICAL TRIAL: NCT03693573
Title: An Open Label, Phase IIIB, Single Arm, Multicenter Safety Study of Atezolizumab in Combination With Bevacizumab in Untreated Locally Advanced or Metastatic Clear Cell or Non-Clear Cell Renal Cell Carcinoma
Brief Title: A Study of Atezolizumab in Combination With Bevacizumab in Untreated Locally Advanced or Metastatic Clear Cell or Non-Clear Cell Renal Cell Carcinoma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: In the context of the ongoing evaluation of our data, we have determined that there is no need to generate additional safety data at this time in the 1L mRCC pa
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO39939
Record Dates: First submitted 2018-09-25; First posted 2018-10-03 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Atezolizumab + Bevacizumab (Experimental): Participants will receive atezolizumab in combination with bevacizumab.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered by intravenous (IV) infusion at a fixed dose of 1200 mg on Day 1 of each 21-day cycle. Administration of study drugs will continue until unacceptable toxicity; loss of clinical benefit as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status; investigator or patient decision to withdraw from therapy; or death (whichever occurs first).
  Other Names: Tecentriq
Drug: Bevacizumab — Bevacizumab will be administered by IV infusion at 15 mg/kg on Day 1 of each 21-day cycle. Administration of study drugs will continue until unacceptable toxicity; loss of clinical benefit as determined by the investigator after an integrated assessment of radiographic and biochemical data, local biopsy results (if available), and clinical status; investigator or patient decision to withdraw from therapy; or death (whichever occurs first).
  Other Names: Avastin

SUMMARY:
Study MO39939 is an open-label, single-arm, multicenter trial in patients with unresectable, locally-advanced or metastatic, clear or non-clear cell renal cell carcinoma (RCC) who have not received prior systemic therapy (who are treatment naïve in either the [neo]adjuvant or advanced/metastatic setting for clear and non-clear cell RCC). The study consists of a Screening Period, a Treatment Period, an End of Treatment Visit occurring approximately 30 days after the last dose of study medication, and a Follow-Up Period of 4 years after last patient enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable, advanced or metastatic RCC with clear cell or non-clear cell histology
* No prior treatment with active or experimental systemic agents for RCC
* Measurable and/or non-measurable but evaluable baseline disease per RECIST v1.1
* Confirmed diagnosis of RCC
* Karnofsky Performance Score (KPS) ≥ 60
* Adequate hematologic and end-organ function
* Patients with asymptomatic CNS metastases are eligible, provided they meet all of the following criteria:

  * Evaluable disease outside the CNS
  * No history of intracranial or spinal cord hemorrhage
  * No evidence of significant vasogenic edema
  * No stereotactic radiation within 7 days or whole-brain radiation or neurosurgical resection within 2 weeks before the start of study treatment
  * Have had a screening CNS radiography ≥ 2 weeks since completion of radiotherapy or surgical resection
* For women of childbearing potential: agreement to remain abstinent or use contraceptive methods, and agreement to refrain from donating eggs
* For men: agreement to remain abstinent or use a condom, and agreement to refrain from donating sperm

Exclusion Criteria:

* Prior treatment for RCC with active or experimental systemic agents, including treatment in the neoadjuvant or adjuvant setting - Confirmed prior treatment with placebo in the (neo)adjuvant setting is allowed
* Radiotherapy ongoing at the time of study entry
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently) - Patients with indwelling catheters are allowed
* Uncontrolled or symptomatic hypercalcemia - Patients who are currently receiving bisphosphonate therapy without current hypercalcemia are eligible
* History of malignancy other than RCC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death, such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer
* Life expectancy of < 12 weeks
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan - History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Active tuberculosis
* Significant renal disorder requiring dialysis
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* Patients with active hepatitis B or hepatitis C
* Current treatment with anti-viral therapy for HBV
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-11 (Estimated); Primary Completion 2021-08-14 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events | Up to 6 years

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 6 years
  OS is defined as the time from enrolment in the study to death from any cause
Progression-Free survival (PFS) | Up to 6 years
  PFS is defined as the time from enrolment in the study to the first occurrence of disease progression or death from any cause, whichever occurs first. PFS will be assessed by the investigator according to RECIST v1.1 and modified RECIST (iRECIST)
Overall Response Rate (ORR) | Up to 6 years
  ORR is defined as the proportion of patients with a best overall response of either complete response (CR) or partial response (PR). ORR will be assessed by the investigator according to RECIST v1.1 and iRECIST.
Disease Control Rate (DCR) | Up to 6 years
  DCR is defined as the sum of the CR, PR and stable disease (SD) rates. DCR will be assessed by the investigator according to RECIST v1.1 and iRECIST.
Duration of Response (DoR) | Up to 6 years
  DoR is defined as the time from first occurrence of a documented response to disease progression or death from any cause, whichever occurs first. DoR will be assessed by the investigator according to RECIST v1.1 and iRECIST.
PD-L1 Expression in Tumor Samples From the Tumor Tissue | At baseline
  Measured retrospectively by immunohistochemistry (IHC).
Change From Baseline in the Single Item (GP5) of the National Comprehensive Cancer Network/Functional Assessment of Cancer Therapy-Kidney Symptom Index 19 (FKSI-19), Version 2 | Before dosing on Day 1 of each cycle, at the End-of-Treatment visit, and at 3, 6, and 9 months after the End-of-Treatment visit. End-of-Treatement visit occurring approximately 30 days after last cycle treatment date. Each cycle is 21 days.
Change From Baseline in MD Anderson Symptom Inventory (MDASI) Core and MDASI-RCC Module | Before dosing on Day 1 of each cycle, at the End-of-Treatment visit, and at 3, 6, and 9 months after the End-of-Treatment visit. End-of-Treatment visit occurring approximately 30 days after last cycle treatment date. Each cycle is 21 days.
Time to Deterioration of Daily Functioning | Before dosing on Day 1 of each cycle, at the End-of-Treatment visit, and at 3, 6, and 9 months after the End-of-Treatment visit. End-of-Treatment visit occurring approximately 30 days after last cycle treatment date. Each cycle is 21 days.
  Time to deterioration of daily functioning is defined as the time from enrolment to first ≥ 2-point increase above baseline in MDASI interference score.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche